CLINICAL TRIAL: NCT04011670
Title: Neuroplastic Alterations of the Motor Cortex by Caffeine: Differences Between Caffeine and Non-caffeine Users and Influence of Vigilance During Stimulation
Brief Title: Neuroplastic Alterations of the Motor Cortex by Caffeine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Walter Paulus, Head of Department for Clinical Neurophysiology, University Medical Center Goettingen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 33/3/19
Record Dates: First submitted 2019-05-21; First posted 2019-07-08 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Cortical Excitability; Brain Stimulation; Caffeine
Keywords: Plasticity; Variability; Non-invasive brain stimulation; Caffeine
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: 15 participants are assigned to caffeine group and another 15 are assigned to placebo group. Then, the participants who were initially in the caffeine group now be in placebo group and those who were in the placebo group were assigned to caffeine group. Finally, all participants received both placebo and caffeine
Who Masked: Participant, Investigator
Masking Description: A statistician prepares a randomization list. Only the pharmacist knows the medication type (caffeine or placebo) and the type of electrical stimulation. The researcher knows only the vigilance conditions (**passive or *active) . An investigator is blinded to the type of electrical stimulation and medication. In addition, all participants are naive to electrical stimulation and do not know if they receive placebo or verum drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine group (Active Comparator): Participants will receive a caffeine tablet and all electrical stimulations in a random order (tACS 140 Hz at 1 mA and sham tACS). Participant's vigilance status will be monitor based on active vigilance condition or passive vigilance condition.
  Interventions: Other: 200 mg caffeine tablet
- Placebo group (Placebo Comparator): Participants will receive a placebo tablet and all electrical stimulations in a random order (tACS 140 Hz at 1 mA and sham tACS). Participant's vigilance status will be monitor based on active vigilance condition or passive vigilance condition.
  Interventions: Other: Non-active tablet

INTERVENTIONS:
Other: 200 mg caffeine tablet — * Transcranial alternating current stimulation (140 Hz tACS) at 1 mA and active vigilance condition
  * Transcranial alternating current stimulation (140 Hz tACS) at 1 mA and passive vigilance condition
  * Transcranial alternating current stimulation (140 Hz tACS) sham and active vigilance condition
  * Transcranial alternating current stimulation (140 Hz tACS) sham and passive vigilance condition
  Arms: Caffeine group
Other: Non-active tablet — * Transcranial alternating current stimulation (140 Hz tACS) at 1 mA and active vigilance condition
  * Transcranial alternating current stimulation (140 Hz tACS) at 1 mA and passive vigilance condition
  * Transcranial alternating current stimulation (140 Hz tACS) sham and active vigilance condition
  * Transcranial alternating current stimulation (140 Hz tACS) sham and passive vigilance condition
  Arms: Placebo group

SUMMARY:
Caffeine is a psychostimulant drug. It acts as a competitive antagonist at adenosine receptors, which modulate cortical excitability as well. In deep brain stimulation (DBS), the production of adenosine following the release of adenosine triphosphate (ATP) explains the reduction of tremor. Binding of adenosine to adenosine A1 receptors suppresses excitatory transmission in the thalamus and hereby reduces both tremor-and DBS-induced side effects. Also, the effect of adenosine was attenuated following the administration of the 8-Cyclopentyl-1,3-dipropylxanthine (DPCPX) adenosine A1 receptor antagonist. Therefore, the presence of a receptor antagonist such as caffeine was suggested to reduce the effectiveness of deep brain stimulation (DBS) in treating tremor and other movement disorders.

Based on this finding, the investigators hypothesize that the antagonistic effect of caffeine can tentatively block the excitatory effects of transcranial alternating current stimulation (tACS). The plasticity effects might differ among caffeine users and non- caffeine users depending on the availability of receptor binding sites.

Apart from that, a major issue in NIBS studies including those studying motor-evoked potentials is the response variability both within and between individuals. The trial to trial variability of motor evoked potentials (MEPs) may be affected by many factors. Inherent to caffeine is its effect on vigilance. In this study, the investigator shall monitor the participant's vigilance by pupillometry to (1) better understand the factors, which might cause variability in transcranial excitability induction studies and (2) to separate the direct pharmacological effect from the indirect attentional effect of caffeine.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female healthy participants between the ages of 18-45.
2. Right-handed (Oldfield 1971).
3. Free willing participation and written, informed consent of all subjects obtained prior to the start of the study.
4. Participant's weight is above 60 kg

Exclusion Criteria:

1. Age < 18 or > 45 years old;
2. Left hand dominant;
3. Evidence of a chronic disease or history with a disorder of the nervous system
4. History of epileptic seizures;
5. Pacemaker or deep brain stimulation;
6. Metal implants in the head region (metal used in the head region, for example, clips after the operation of an intracerebral aneurysm (vessel sacking in the region of the brain vessels), implantation of an artificial auditory canal);
7. Cerebral trauma with loss of consciousness in prehistory;
8. Existence of a serious internal (internal organs) or psychiatric (mental illness)
9. Alcohol, medication or drug addiction;
10. Receptive or global aphasia (disturbance of speech comprehension or additionally of speech);
11. Participation in another scientific or clinical study within the last 4 weeks;
12. Pregnancy
13. Breastfeeding
14. Intolerance to caffeine or coffee products
15. Participant who has abnormal heart activity from an electrocardiography (ECG) finding
16. Weight is less than 60 kg

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Neuroplastic changes of the cortical areas | Baseline (pre-measurement), immediately after intervention, 5 minutes, 10 minutes, 15 minutes, 20 minutes, 25 minutes, 30 minutes
  Motor cortex plasticity is measured from the changes in the amplitude of the motor evoked potentials (MEPs) at different time points. Transcranial magnetic stimulation (TMS) will be used to measure MEP amplitudes.
The influence of vigilance during stimulation | 10 minutes
  Participant's level of vigilance is monitored from pupil diameter and pupil unrest index (PUI) using pupillometer. This measurement is carried out during 10 minutes of transcranial alternating current stimulation (tACS)

SECONDARY OUTCOMES:
Genetic polymorphism | 1 year
  Brain-derived neurotrophic factor (BDNF) gene polymorphisms on cortical plasticity

CONTACTS AND LOCATIONS:
Overall Officials: Walter Paulus, Principal Investigator — University Medical Center Goettingen, Goettingen
Locations (1):
- Prof. Dr. Walter Paulus, Goettigen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Antal A, Chaieb L, Moliadze V, Monte-Silva K, Poreisz C, Thirugnanasambandam N, Nitsche MA, Shoukier M, Ludwig H, Paulus W. Brain-derived neurotrophic factor (BDNF) gene polymorphisms shape cortical plasticity in humans. Brain Stimul. 2010 Oct;3(4):230-7. doi: 10.1016/j.brs.2009.12.003. Epub 2010 Jan 14. PMID 20965453
- [Background] Biabani M, Farrell M, Zoghi M, Egan G, Jaberzadeh S. The minimal number of TMS trials required for the reliable assessment of corticospinal excitability, short interval intracortical inhibition, and intracortical facilitation. Neurosci Lett. 2018 May 1;674:94-100. doi: 10.1016/j.neulet.2018.03.026. Epub 2018 Mar 15. PMID 29551425
- [Background] Cappelletti S, Piacentino D, Sani G, Aromatario M. Caffeine: cognitive and physical performance enhancer or psychoactive drug? Curr Neuropharmacol. 2015 Jan;13(1):71-88. doi: 10.2174/1570159X13666141210215655. PMID 26074744
- [Background] Cappelletti S, Piacentino D, Fineschi V, Frati P, Cipolloni L, Aromatario M. Caffeine-Related Deaths: Manner of Deaths and Categories at Risk. Nutrients. 2018 May 14;10(5):611. doi: 10.3390/nu10050611. PMID 29757951
- [Background] Cavaleri R, Schabrun SM, Chipchase LS. The number of stimuli required to reliably assess corticomotor excitability and primary motor cortical representations using transcranial magnetic stimulation (TMS): a systematic review and meta-analysis. Syst Rev. 2017 Mar 6;6(1):48. doi: 10.1186/s13643-017-0440-8. PMID 28264713
- [Background] Cuypers K, Thijs H, Meesen RL. Optimization of the transcranial magnetic stimulation protocol by defining a reliable estimate for corticospinal excitability. PLoS One. 2014 Jan 24;9(1):e86380. doi: 10.1371/journal.pone.0086380. eCollection 2014. PMID 24475111
- [Background] Feurra M, Paulus W, Walsh V, Kanai R. Frequency specific modulation of human somatosensory cortex. Front Psychol. 2011 Feb 2;2:13. doi: 10.3389/fpsyg.2011.00013. eCollection 2011. PMID 21713181
- [Background] Goldsworthy MR, Hordacre B, Ridding MC. Minimum number of trials required for within- and between-session reliability of TMS measures of corticospinal excitability. Neuroscience. 2016 Apr 21;320:205-9. doi: 10.1016/j.neuroscience.2016.02.012. Epub 2016 Feb 9. PMID 26872998
- [Background] Hanajima R, Tanaka N, Tsutsumi R, Shirota Y, Shimizu T, Terao Y, Ugawa Y. Effect of caffeine on long-term potentiation-like effects induced by quadripulse transcranial magnetic stimulation. Exp Brain Res. 2019 Mar;237(3):647-651. doi: 10.1007/s00221-018-5450-9. Epub 2018 Dec 10. PMID 30535949
- [Background] Higdon JV, Frei B. Coffee and health: a review of recent human research. Crit Rev Food Sci Nutr. 2006;46(2):101-23. doi: 10.1080/10408390500400009. PMID 16507475
- [Background] Karabanov A, Ziemann U, Hamada M, George MS, Quartarone A, Classen J, Massimini M, Rothwell J, Siebner HR. Consensus Paper: Probing Homeostatic Plasticity of Human Cortex With Non-invasive Transcranial Brain Stimulation. Brain Stimul. 2015 May-Jun;8(3):442-54. doi: 10.1016/j.brs.2015.01.404. Epub 2015 Apr 1. PMID 26050599
- [Background] Di Lazzaro V, Pellegrino G, Di Pino G, Corbetto M, Ranieri F, Brunelli N, Paolucci M, Bucossi S, Ventriglia MC, Brown P, Capone F. Val66Met BDNF gene polymorphism influences human motor cortex plasticity in acute stroke. Brain Stimul. 2015 Jan-Feb;8(1):92-6. doi: 10.1016/j.brs.2014.08.006. Epub 2014 Aug 23. PMID 25241287
- [Background] Lewis GN, Signal N, Taylor D. Reliability of lower limb motor evoked potentials in stroke and healthy populations: how many responses are needed? Clin Neurophysiol. 2014 Apr;125(4):748-754. doi: 10.1016/j.clinph.2013.07.029. Epub 2013 Oct 5. PMID 24103535
- [Background] Marquez-Ruiz J, Leal-Campanario R, Sanchez-Campusano R, Molaee-Ardekani B, Wendling F, Miranda PC, Ruffini G, Gruart A, Delgado-Garcia JM. Transcranial direct-current stimulation modulates synaptic mechanisms involved in associative learning in behaving rabbits. Proc Natl Acad Sci U S A. 2012 Apr 24;109(17):6710-5. doi: 10.1073/pnas.1121147109. Epub 2012 Apr 9. PMID 22493252
- [Background] Moliadze V, Antal A, Paulus W. Boosting brain excitability by transcranial high frequency stimulation in the ripple range. J Physiol. 2010 Dec 15;588(Pt 24):4891-904. doi: 10.1113/jphysiol.2010.196998. PMID 20962008
- [Background] Moliadze V, Antal A, Paulus W. Electrode-distance dependent after-effects of transcranial direct and random noise stimulation with extracephalic reference electrodes. Clin Neurophysiol. 2010 Dec;121(12):2165-71. doi: 10.1016/j.clinph.2010.04.033. Epub 2010 Jun 15. PMID 20554472
- [Background] Moliadze V, Atalay D, Antal A, Paulus W. Close to threshold transcranial electrical stimulation preferentially activates inhibitory networks before switching to excitation with higher intensities. Brain Stimul. 2012 Oct;5(4):505-11. doi: 10.1016/j.brs.2011.11.004. Epub 2012 Feb 22. PMID 22445135
- [Background] Muller-Dahlhaus F, Ziemann U. Metaplasticity in human cortex. Neuroscientist. 2015 Apr;21(2):185-202. doi: 10.1177/1073858414526645. Epub 2014 Mar 11. PMID 24620008
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Polania R, Nitsche MA, Korman C, Batsikadze G, Paulus W. The importance of timing in segregated theta phase-coupling for cognitive performance. Curr Biol. 2012 Jul 24;22(14):1314-8. doi: 10.1016/j.cub.2012.05.021. Epub 2012 Jun 7. PMID 22683259
- [Background] Ridding MC, Ziemann U. Determinants of the induction of cortical plasticity by non-invasive brain stimulation in healthy subjects. J Physiol. 2010 Jul 1;588(Pt 13):2291-304. doi: 10.1113/jphysiol.2010.190314. Epub 2010 May 17. PMID 20478978
- [Background] Robertson D, Wade D, Workman R, Woosley RL, Oates JA. Tolerance to the humoral and hemodynamic effects of caffeine in man. J Clin Invest. 1981 Apr;67(4):1111-7. doi: 10.1172/jci110124. PMID 7009653
- [Background] Stefan K, Kunesch E, Cohen LG, Benecke R, Classen J. Induction of plasticity in the human motor cortex by paired associative stimulation. Brain. 2000 Mar;123 Pt 3:572-84. doi: 10.1093/brain/123.3.572. PMID 10686179
- [Background] Stefan K, Kunesch E, Benecke R, Cohen LG, Classen J. Mechanisms of enhancement of human motor cortex excitability induced by interventional paired associative stimulation. J Physiol. 2002 Sep 1;543(Pt 2):699-708. doi: 10.1113/jphysiol.2002.023317. PMID 12205201
- [Background] Zaehle T, Rach S, Herrmann CS. Transcranial alternating current stimulation enhances individual alpha activity in human EEG. PLoS One. 2010 Nov 1;5(11):e13766. doi: 10.1371/journal.pone.0013766. PMID 21072168
- [Derived] Zulkifly MFM, Merkohitaj O, Brockmoller J, Paulus W. Confounding effects of caffeine on neuroplasticity induced by transcranial alternating current stimulation and paired associative stimulation. Clin Neurophysiol. 2021 Jun;132(6):1367-1379. doi: 10.1016/j.clinph.2021.01.024. Epub 2021 Mar 10. PMID 33762129
- [Derived] Zulkifly MFM, Merkohitaj O, Paulus W, Brockmoller J. The roles of caffeine and corticosteroids in modulating cortical excitability after paired associative stimulation (PAS) and transcranial alternating current stimulation (tACS) in caffeine-naive and caffeine-adapted subjects. Psychoneuroendocrinology. 2021 May;127:105201. doi: 10.1016/j.psyneuen.2021.105201. Epub 2021 Mar 15. PMID 33740589